CLINICAL TRIAL: NCT07325708
Title: Clinical Evaluation of System for Bionic Arm Gesture Control (CYBORG)
Brief Title: Evaluation of the Phantom X Implantable EMG Sensor System for Myoelectric Prosthesis Control
Acronym: CYBORG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phantom Neuro Inc. (Industry)
Collaborators: Cabrini Health, Melbourne, Australia (Unknown); ProMotion Prosthetics, Moorabbin, Australia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PN03
Record Dates: First submitted 2025-12-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Upper Limb Amputation Below Elbow (Injury); Wrist Disarticulation; Transradial Amputation
Keywords: Upper limb amputation; Prosthesis; Myoelectric
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Phantom X (Experimental)
  Interventions: Device: Phantom X multielectrode EMG sensor array implant for upper limb prosthesis control

INTERVENTIONS:
Device: Phantom X multielectrode EMG sensor array implant for upper limb prosthesis control — Participants receive the Phantom X implantable EMG sensor array and telemetry module to enable myoelectric control of an upper-limb prosthesis.

SUMMARY:
The CYBORG Study is a first-in-human clinical investigation evaluating the safety and performance of the Phantom X System, an implantable electromyography (EMG) sensor array designed to provide control of upper-limb prostheses. The study will assess surgical feasibility, device function, signal quality, and the system's ability to support intuitive prosthetic control during functional tasks. Participants will undergo implantation of the Phantom X sensors and complete a series of in-clinic visits to assess functional performance of the Phantom X system. Patient-reported outcomes will also be collected at various timepoints.

DETAILED DESCRIPTION:
This early-feasibility study will evaluate the safety and functional performance of the Phantom X Implantable EMG Sensor System in individuals with unilateral transradial amputation and wrist disarticulation. The system consists of an implanted EMG sensor array, an implanted telemetry module, and an external wearable interface that provides real-time muscle signals to a myoelectric prosthesis.

The study follows a prospective, single-arm, open label design. Participants will undergo surgical implantation followed by device activation, calibration, and integration with a compatible prosthetic hand. Study procedures include periodic assessments of EMG signal quality, standardized functional assessments, and patient reported outcomes including quality of life measures and user experience. Safety will be monitored through adverse-event reporting and system performance checks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a unilateral upper-limb difference (congenital or acquired) at the transradial or wrist level.
2. The patient currently uses a myoelectric prosthesis or is deemed a suitable candidate for fitting with a myoelectric prosthesis.
3. Patient is a suitable candidate for the implantation of the Phantom X sensor array as assessed by the implanting physician.
4. Patient is at least 18 years old and can provide written informed consent.
5. Patient is willing to comply with study protocol and make required study visits.
6. Patient received amputation ≥ 12 months prior to consent.

Exclusion Criteria:

1. Patient has a significant cognitive deficit resulting in inability to follow study directions.
2. Patient has a neuro-muscular deficit and is unable to initiate substantial muscle contraction in the residual limb as determined by the implanting physician or investigator.
3. Patient has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
4. The patient has a planned medical procedure (e.g., surgery) during the study period that could interfere with compliance with study visits or assessments.
5. Patient has an allergy to anesthesia or other medication used for sedation in the study.
6. Patient has an active implantable device (e.g. cardiac pacemaker, neuromodulation device) that can potentially interfere with the performance of Phantom X system.
7. Patient may require an MRI during the study duration.
8. Implantation of the device poses a health risk to the patient as determined by the implanting physician.
9. Women who are breastfeeding, currently pregnant or planning to become pregnant during the duration of the study or have a positive urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety of Phantom X system during the implantation procedure, peri-procedurally, and 9 weeks thereafter | 9 weeks
  Safety is characterized by collecting device and procedure related adverse events during device implantation and 9-week study follow-up.
Functionality of Phantom X system using standardized Assessment of Capacity for Myoelectric Control (ACMC) instrument | 9 weeks
  Average and standard deviation of ACMC scores will be computed for all participants
Functionality of Phantom X system using standardized Targeted Box and Blocks Test (tBBT) instrument | 9 weeks
  Average and standard deviation of tBBT scores will be computed for all participants

SECONDARY OUTCOMES:
Safety of Phantom X system during the implantation procedure, peri-procedurally, and 21 weeks thereafter | 21 weeks
  Safety is characterized by collecting device and procedure related adverse events during device implantation and 21-week study follow-up.
Functionality of Phantom X system using standardized Assessment of Capacity for Myoelectric Control (ACMC) instrument | 21 weeks
  Average and standard deviation of ACMC scores will be computed for all participants
Functionality of Phantom X system using standardized Targeted Box and Blocks Test (tBBT) instrument | 21 weeks
  Average and standard deviation of tBBT scores will be computed for all participants
Phantom X Signal-to-Noise Ratio (SNR) | 9 weeks and 21 weeks
  Characterize signal-to-noise ratio (SNR) of electromyography (EMG) signals obtained using Phantom X system. Average and standard deviation of SNR for all participants will be computed
Phantom X algorithm gesture accuracy | 9 weeks and 21 weeks
  Classification accuracy of the Phantom X algorithm will be computed based on the number of correctly and incorrectly classified gestures and reported as a percentage
Phantom X at-home wear duration | 9 weeks and 21 weeks
  Average and standard deviation of at-home prosthesis wear duration for all participants will be computed
At-home limb usage pattern using Inertial Measurement Unit (IMU) data | 9 weeks and 21 weeks
  Active and inactive durations in hours per day for each limb will be computed for each participant
Prosthesis control resolution | 9 weeks and 21 weeks
  Resolution of Phantom X control system for controlling a myoelectric hand prosthesis will be characterized using Myoelectric Control Resolution Assessment (MCRA) instrument
Number of system recalibration events | 9 weeks and 21 weeks
  Number of Phantom X recalibrations per participant will be collected and used to compute average and standard deviation of recalibration events for all participants
User Satisfaction | 9 weeks and 21 weeks
  User Satisfaction with Phantom X system is characterized using following three standardized instruments: modified version of Orthotics Prosthetics User Survey (mOPUS, range: 0-100, Higher score is better), 5-level Quality of Life questionnaire (EQ-5D-5L, Higher score is better), Canadian Occupational Performance Measure (COPM, range:1-10, Higher score is better), and a study User Satisfaction Survey.
Robustness of Phantom X system | 9 weeks and 21 weeks
  Robustness of Phantom X system is characterized by recording problematic activities of daily living (REC-ADL) that participants have problem performing with their baseline myoelectric control system.
Phantom X ease of use | 9 weeks and 21 weeks
  Ease of use and intuitiveness of Phantom X system is characterized using NASA-Task Load Index (NASA-TLX) instrument.
Phantom Limb Pain | 9 weeks and 21 weeks
  Change in phantom limb pain is characterized post implant and compared with baseline using Questionnaire for Post-Amputation Pain (Q-PAP).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lo, MBBS, FRACS, BSc (Hons), Principal Investigator — Cabrini Private Hospital, Malvern, Australia
Locations (2):
- Australia (2):
  - Cabrini Health Ltd, Malvern, Victoria
  - ProMotion Prosthetics Pty Ltd, Moorabbin, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
We may not share IPD because of concerns about protecting participants' privacy and confidentiality. Even though our participant data would be de-identified, there is a risk (especially with sensitive, rare, or detailed clinical data as would be the case for amputees in our study) that the individuals could be re-identified. Maintaining confidentiality and minimizing potential harm to participants may outweigh the benefits of data sharing.